CLINICAL TRIAL: NCT03182127
Title: Role of Magnetic Resonance Imaging in Evaluation of Non-traumatic Causes of Painful Elbow Joint
Brief Title: Role of MRI in Evaluation of Non-traumatic Causes of Painful Elbow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara gamal mohammad, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRI IN ELBOW JOINT
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Elbow Disease
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one Group (Other): Magnetic resonance imaging and ultrasound will be done for all patient
  Interventions: Radiation: Magnetic resonance imaging; Device: Ultrasound

INTERVENTIONS:
Radiation: Magnetic resonance imaging — MRI of the elbow is performed in either the supine or prone position A high-resolution surface coil is essential in order to obtain high-quality images . Elbow MRI scanning protocols consist of a combination of T1-weighted and fat-suppressed T2- or proton density-weighted images obtained in the axial, coronal oblique, and sagittal oblique imaging planes. Axial images should extend from the distal humeral diaphysis to the level of the bicipital tuberosity of the radius. From the axial images, coronal oblique images should be prescribed parallel to a line drawn through the centre of the humeral epicondyles, with sagittal oblique images prescribed perpendicular to this. Additional sequences may be helpful in certain circumstances; .
Device: Ultrasound — ultrasound is performed by patient in supine or setting position,applied superficial probe , 2D image and color doppler if indicated.

SUMMARY:
• Elbow pain is any type of pain that comes from structures in the elbow joint and/or in structures adjacent to the elbow joint. elbow is a complex joint; it allows to both extension and flexion, as well as rotation hand and forearm. Since most movements are a combination of these actions, Elbow pain is often caused by overuse, but in general, elbow joint is much less prone to wear-and-tear damage than are many other joints. The causes of elbow pain are numerous. Most elbow pain is due to overuse or strain on the elbow joint components, but some causes are due to trauma, infection, and/or autoimmune processes and neoplasm. Risk factors for elbow pain are numerous and range from engaging in repetitive activities and participation in sports to those associated with infection, trauma, and rheumatoid arthritis. Other adjacent structures associated with elbow pain include the shoulder, upper arm, forearm, and wrist and hand joints.

DETAILED DESCRIPTION:
* Health-care professionals diagnose elbow pain mainly by a patient's history and physical exam. Radiologic techniques such as X-ray ,US,CT and MRI are often used to delineate the elbow structures involved. Conventional radiography remains an essential initial test in the evaluation of the elbow and its disorders. One must be familiar with the pertinent anatomy, early developmental changes, and the biomechanics of this complex joint to appreciate subtle injury patterns and articular disorders. In some cases, radiographic imaging will point to the need for further evaluation with CT, MR, or sonographic imaging High-resolution ultrasound is well suited for evaluating the elbow. Ultrasound is growing in popularity and fast becoming another modality that the radiologist can use to help diagnose elbow pathology. ultrasound offers focused and real-time high-resolution imaging of tendons, ligaments, and nerve structures. Its advantages include the use of safe nonionizing radiation, accessibility, and cost effectiveness. Ultrasound is also useful in therapeutic guided injections for its multiplanar capability and clear visualization of major vessels and nerves.
* MR imaging provides clinically useful information in assessing the elbow joint. Superior depiction of muscles, ligaments, and tendons as well as the ability to visualize nerves, bone marrow, and hyaline cartilage directly are advantages of MR imaging relative to conventional imaging techniques. These features of MR imaging may help to establish the cause of elbow pain by accurately depicting the presence and extent of bone and soft-tissue pathology. Ongoing improvements in surface coil design and newer pulse sequences have resulted in higher quality MR images of the elbow that can be obtained more rapidly. This is especially important in MR as the imaging tool that shows a highest soft tissue resolution among other imaging techniques. Recent clinical experience has shown the utility of MR imaging in detecting and characterizing disorders of the elbow in a a noninvasive fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of elbow pain not related by trauma.
2. Cases with self-reported history of overuse, infection, autoimmune disease, bleeding tendency and neoplasm of bone, joint, soft tissue at elbow.

Exclusion Criteria:

1. Recent acute traumatic cases.
2. Cases not fulfilling MRI criteria(contraindicated for MRI): metal implant (pacemaker, artificial valve prosthesis ,implantable cardiovascular defibrillator, nerve simulator, intro-ocular implant, cochlear implants, arterial clips, bullets or metal fragments, swan-guns catheter).
3. Pregnancy and breast milk feeding.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with non-traumatic painful elbow is diagnosed by MRI Using sensitivity, specificity and accuracy tests which used for . | 6 Months
  :46 cases, is calculated using the Open Epi software programme, version 2.3.1. previous study reported the expected rate 40%. estimated the increase into 40% (80%). using two sided chi-square (x-2) test with alpha (95%). total sample size of at least (46) using 80% power will be needed (odd ratio=0.17). assuming a rate of drop-out of (10%), so, will include (46) cases.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gamal, Residant, Principal Investigator — Assiut University
Locations (1):
- Assiut, Assiut,Egypt, Egypt

REFERENCES:
- [Background] Read PJ, Morrison WB. Imaging Injuries in Throwing Sports Beyond the Typical Shoulder and Elbow Pathologies. Radiol Clin North Am. 2016 Sep;54(5):857-64. doi: 10.1016/j.rcl.2016.05.001. PMID 27545424